CLINICAL TRIAL: NCT03232827
Title: The Impact of Waterpipe Tobacco Flavors on Waterpipe Smoking Intentions, Perceptions, Patterns, and Toxicant Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Virginia Commonwealth University (Other); American University of Beirut Medical Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R03DA041928-01A1 (NIH); 1R03DA041928-01A1 (NIH)
Record Dates: First submitted 2017-06-22; First posted 2017-07-28 (Actual); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Smoking, Hookah; Waterpipe Smoking
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flavored-sweetened (Active Comparator): Flavored-sweetened (FS) WP tobacco will be associated with longer and more frequent puffing resulting in the greatest overall levels of smoke inhalation (mL of smoke inhaled), highest abuse potential, and greatest levels of exposure to nicotine and carbon monoxide (CO). , followed by unflavored-sweetened WP, and lastly unflavored-very low sweetened WP. (H1d) A majority of WP smokers will report having initiated WP smoking with flavored-sweetened tobacco and report flavoring as an important reason for trying WP.
  Interventions: Behavioral: Flavored-Sweetened Waterpipe Tobacco
- Unflavored-sweetened (Active Comparator): Unflavored-sweetened (US) WP will be associated with the second longest and slightly less frequent puffing than FS resulting in the second greatest overall levels of smoke inhalation (mL of smoke inhaled), abuse potential, and levels of exposure to nicotine and carbon monoxide (CO).
  Interventions: Behavioral: Unflavored-sweetened waterpipe tobacco
- Unflavored very low sweetened (Active Comparator): Unflavored-very low sweetened (UU) WP will be associated with the shortest and the least frequent puffing resulting in the least overall levels of smoke inhalation (mL of smoke inhaled), abuse potential, and levels of exposure to nicotine and carbon monoxide (CO).
  Interventions: Behavioral: Unflavored-very low sweetened waterpipe tobacco
- Flavored-very low sweetened waterpipe (Active Comparator): Flavored-very low sweetened WP will be associated with the third longest and slightly less frequent puffing than US resulting in the third greatest overall levels of smoke inhalation (mL of smoke inhaled), abuse potential, and levels of exposure to nicotine and carbon monoxide (CO).
  Interventions: Behavioral: Flavored-very low sweetened waterpipe

INTERVENTIONS:
Behavioral: Flavored-Sweetened Waterpipe Tobacco — Pre-weighed flavored-sweetened waterpipe tobacco will be prepared.
  Arms: Flavored-sweetened
Behavioral: Unflavored-sweetened waterpipe tobacco — Pre-weighed unflavored-sweetened waterpipe tobacco will be prepared.
  Arms: Unflavored-sweetened
Behavioral: Unflavored-very low sweetened waterpipe tobacco — Pre-weighed unflavored-very low sweetened waterpipe tobacco will be prepared.
  Arms: Unflavored very low sweetened
Behavioral: Flavored-very low sweetened waterpipe — Pre-weighed flavored-very low sweetened waterpipe tobacco will be prepared.
  Arms: Flavored-very low sweetened waterpipe

SUMMARY:
The overall aim of the current study is to determine if flavorings contribute to the initiation and maintenance of waterpipe (WP) smoking and also influence how a WP is smoked, which has implications for both risk of dependence but also smokers' level of exposure to tobacco-related toxicants. A total of 94 current WP smokers (47 low dependent, 47 high dependent) will be recruited. Based on our team's previous studies we conservatively assume a 20% attrition rate; thus, we will need to recruit 94 participants to have 76 complete all four sessions. Consistent with other laboratory studies of waterpipe smoking, participants who meet the following eligibility criteria will be asked to take part in the study.

DETAILED DESCRIPTION:
After completing the initial screening by phone, participants will be informed of the study procedures and invited to the lab to complete three WP smoking sessions. Participants will perform exhaled carbon monoxide testing (eCO< 10ppm) and confirm that they have not used any nicotine/tobacco/marijuana products over the last 12 hours. Pregnancy exclusion will also be confirmed with a urine test, and pregnancy tests will be completed at each visit throughout the study. Participants will be randomized and complete study procedures in self-selected dyads. The sessions will be counterbalanced and include: 1) smoking preferred flavored-sweetened WP tobacco, 2) smoking unflavored-sweetened WP tobacco, and 3) smoking unflavored-very low sweetened WP tobacco. Participants will complete all three study visits in the laboratory. Pre-session abstinence from tobacco for at least 12 hours will be mandatory for all participants. Abstinence will be confirmed via participant self-report and an exhaled carbon monoxide monitor (< 20 ppm) for tobacco use. Participant dyads will smoke hookah ad libitum for up to 1 hour. This procedure will be completed for all visits. Participants will also complete a minimum 48-hour washout period between sessions.

Participants will not be allowed to eat, drink or use their phone during the session. Initially, one piece of charcoal will be lit and placed on top of the foil. Our preliminary studies, as well as other WP laboratory trials, indicate that one piece of charcoal will not be sufficient for one WP session; thus, participants will be provided additional pre-weighed pieces to use as they wish. Use of additional charcoal will be recorded. Participants will smoke ad libitum and a WP puff topography device will discretely record smoking behavior throughout the session, including puff duration, number of puffs, puff volume, puff flow rate, and time between puffs. Blood samples (15mL per sample) and eCO will be collected immediately pre- and post-waterpipe session. Self-report measures will be administered.

ELIGIBILITY:
Inclusion Criteria:

* current water pipe smoker for at least the past 6 months
* smoke water pipe at least 3 times in the last 6 months
* Lebanese Waterpipe Dependence Scale-11 (LWDS-11) score of ≤9 (Low Dependence) or ≥10 (High Dependence)
* between 18-50 years old
* willing to provide informed consent
* abstain from all tobacco, nicotine, and marijuana use for at least 12 hours prior to each of the three sessions

Exclusion Criteria:

* self-reported diagnosis of lung disease including asthma, cystic fibrosis, or chronic obstructive pulmonary disease
* currently pregnant, planning to become pregnant, or breastfeeding
* history of cardiac event or distress within the last 3 months
* any use of other illicit drugs during the last 30 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Wagener, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center Tobacco Research Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 207 individuals were identified as eligible for study participation. Study personnel contacted the individuals by telephone to schedule their initial visit. 91 were consented and enrolled.
Pre-assignment Details: Subjects who were eligible & presented to initial visit 12 hour tobacco abstinent were randomized. Subjects were randomized to 1 of 36 session sequences & completed up to four smoking sessions. 2 subjects were not nicotine abstinent at their initial visit, were rescheduled & lost to follow-up.
Groups:
- All Interventions: Participants will be randomized and complete study procedures in self-selected dyads. The sessions will be counterbalanced and include: 1) smoking preferred flavored-sweetened WP tobacco 2) smoking unflavored-sweetened WP Tobacco and 3) smoking preferred flavored-very low sweetened WP tobacco and 4) smoking unflavored-very low sweetened WP tobacco. Participants will complete all four study visits in the laboratory. Pre-session abstinence from tobacco for at least 12 hours will be mandatory for all participants. Abstinence will be confirmed via participant self-report and an exhaled carbon monoxide monitor (< 20 ppm) for tobacco use. Participant dyads will first complete a 10-minute puffing session separated by 30-second intervals with the prepared hookah and then smoke ad libitum for up to 1 hour. This procedure will be completed for all visits. Participants will also complete a minimum 48-hour washout period between sessions.
Period: Flavored-sweetened (FS)
Arm/Group | All Interventions
Started | 80
Completed | 80
Not Completed | 0
Period: Unflavored-sweetened (US)
Arm/Group | All Interventions
Started | 86
Completed | 86
Not Completed | 0
Period: Unflavored-very Low Sweetened (UU)
Arm/Group | All Interventions
Started | 66
Completed | 66
Not Completed | 0
Period: Flavored-very Low Sweetened
Arm/Group | All Interventions
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants completed up to 4 smoking sessions and were randomized to 1 of 36 session sequences: 1) FS - UU - US, 2) UU - FS - US, 3) US - UU - FS, 4) FS - US - UU, 5) US - FS - UU, 6) UU - US - FS, 7) UU - FU - US - FS, 8) UU - FU - FS - US, 9) UU - US - FS - FU, 10) UU - US - FU - FS, 11) UU - FS - US - FU, 12) UU - FS - FU - US, 13) FU - UU - US - FS, 14) FU - UU - FS - US, 15) FU - US - FS - UU, 16) FU - US - UU - FS, 17) FU - FS - UU - US, 18) FU - FS - US - UU, 19) US - UU - FU - FS, 20) US - UU - FS - FU, 21) US - FU - UU - FS, 22) US - FU - FS - UU, 23) US - FS - UU - FU, 24) US - FS - FU - UU, 25) FS - UU - FU - US, 26) FS - UU - US - FU, 27) FS - FU - UU - US, 28) FS - FU - US - UU, 29) FS - US - FU - UU, 30) FS - US - UU - FU, 31) UU - FU - FS - US, 32) FS - UU - FU - US, 33) FU - FS - US - UU, 34) US - UU - FS - FU, 35) FU - US - UU - FS, 36) UU - US - FU - FS. A fourth arm (FU) was added to the study one month after the study started.
Arm/Group | All Study Participants
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.98 (5.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 48
  More than one race | 10
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 89
Waterpipe smoking days per month [Mean (Standard Deviation); unit: Days] | 6.5 (8.3)
Waterpipe dependence [Count of Participants; unit: Participants] — WP dependence will be measured using the Lebanese Waterpipe Dependence Scale-11. ≤9 (Low Dependence) or ≥10 (High Dependence). This validated scale is correlated significantly with nicotine exposure, CO, and WP use frequency. The 11 scale items were summed to calculate the total WP dependence score. The cutoffs for low vs high dependence are as follows: ≤9 (Low Dependence) or ≥10 (High Dependence).
  Participants
    Low Dependence | 50
    High Dependence | 39

OUTCOME MEASURES:

1. Primary Outcome: Level of Smoke Inhalation Measured by Topography Device
Description: Participants will complete one ad-lib puffing session at each visit. Levels of smoke inhalation will be measured throughout each ad-lib puffing session. Flavored-sweetened WP tobacco will be associated with longer and more frequent puffing resulting in the greatest overall levels of smoke inhalation (mL of smoke inhaled).
Time Frame: 6 months
Population: 1 participant was not included in analysis due to self-withdraw. Participants who completed one or more of the individual intervention visits were included.
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Flavored-sweetened | Unflavored-sweetened | Unflavored Very Low Sweetened | Flavored-very Low Sweetened Waterpipe
Number analyzed (Participants) | 80 | 86 | 66 | 66
Liters | 50.96 (5.46) | 77.79 (5.89) | 63.17 (5.87) | 51.60 (4.63)

2. Secondary Outcome: Levels of Smoke Inhalation Between High vs. Low Dependent WP
Description: Waterpipe dependence for participants will be determined at baseline. Participants will complete one ad-lib puffing session at each visit. Levels of smoke inhalation will be measured throughout each ad-lib puffing session. Flavored-sweetened WP tobacco will be associated with longer and more frequent puffing resulting in the greatest overall levels of smoke inhalation (mL of smoke inhaled). Compared to high dependence users smoking unflavored WP tobacco, low dependence users will show greater declines in (H2a) puff frequency and duration resulting in lower levels of smoke inhalation
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Flavored-sweetened | Unflavored-sweetened | Unflavored Very Low Sweetened | Flavored-very Low Sweetened Waterpipe
Number analyzed (Participants) | 80 | 86 | 66 | 66
Liters
  Low Dependence: number analyzed (Participants) | 48 | 48 | 41 | 40
  Low Dependence | 42.18 (5.02) | 55.85 (5.84) | 46.18 (6.03) | 39.43 (4.54)
  High Dependence: number analyzed (Participants) | 32 | 38 | 25 | 26
  High Dependence | 32.15 (6.26) | 57.31 (6.95) | 51.07 (7.26) | 33.96 (5.01)

ADVERSE EVENTS:
Time Frame: Participants were monitored over the 6 months they were in the study. Adverse event information was collected and assessed at each visit.
Groups:
- Flavored Sweetened: Flavored-sweetened (FS) WP tobacco will be associated with longer and more frequent puffing resulting in the greatest overall levels of smoke inhalation (mL of smoke inhaled), highest abuse potential, and greatest levels of exposure to nicotine and carbon monoxide (CO). , followed by unflavored-sweetened WP, and lastly unflavored-very low sweetened WP. (H1d) A majority of WP smokers will report having initiated WP smoking with flavored-sweetened tobacco and report flavoring as an important reason for trying WP.
- Unflavored Sweetened: Unflavored-sweetened (US) WP will be associated with the second longest and slightly less frequent puffing than FS resulting in the second greatest overall levels of smoke inhalation (mL of smoke inhaled), abuse potential, and levels of exposure to nicotine and carbon monoxide (CO).
  Unflavored-sweetened waterpipe tobacco: Pre-weighed unflavored-sweetened waterpipe tobacco will be prepared.
Arm/Group | Flavored Sweetened | Unflavored Sweetened | Unflavored Very Low Sweetened | Flavored-very Low Sweetened Waterpipe
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/86 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/86 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/80 | 0/86 | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03232827/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03232827/Prot_SAP_001.pdf